CLINICAL TRIAL: NCT06212089
Title: Phase II Clinical Study of TR-012001 in Japanese Patients With Parkinson's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SNLD, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TR-012001-PD201
Record Dates: First submitted 2023-12-21; First posted 2024-01-18 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TR-012001 (Experimental): Single dose of TR-012001
  Interventions: Drug: TR-012001
- Placebo (Other): Single dose of placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: TR-012001 — A single dose of TR-012001 will be administered.
  Arms: TR-012001
Other: Placebo — A single dose of placebo will be administered.
  Arms: Placebo

SUMMARY:
The purpose of this study to evaluate the safety and pharmacokinetics of TR-012001 in patients with Parkinson's disease when TR-012001 or placebo is administered.

ELIGIBILITY:
Inclusion Criteria:

* Japanese males and females aged 30 years or older at the time of informed consent.
* Patients diagnosed with idiopathic Parkinson's disease according to the UKPDS Brain Bank Parkinson's disease diagnostic criteria.
* Patients with Parkinson's disease stage 2-4 on the modified Hoehn & Yahr Scale in the "ON state".
* Patients who are taking levodopa-containing drugs* three times or more per day, with a daily dosage of 300 mg or more of levodopa.

  *Levodopa-containing drugs: Levodopa/dopa decarboxylase inhibitor (DCI) combination drugs; DCI can be either carbidopa or benserazide.
* Patients who can maintain a fixed dosage and administration of levodopa-containing drugs and other antiparkinsonian drugs (only for patients taking medication) after obtaining informed consent until the end of the study.
* Patients who are found to be OFF in their daily life by patient evaluation.
* Females of childbearing potential** or males with female partners of childbearing potential** who agree to practice adequate contraception on a daily basis from the time consent is obtained until the end of the study.

  **Female (partners) of childbearing potential: Women who have not confirmed menopause (no menstruation for 52 weeks or more counting from the start of the last menstrual period).
* Patients who are fully informed about the purpose and contents of this study before the start of screening, who understand the contents of the informed consent form, and who can sign their own will.

Exclusion Criteria:

* Patients with non-idiopathic Parkinson's disease [atypical Parkinson's disease, secondary (acquired or symptomatic) Parkinson's disease, Parkinson's plus syndrome, etc.].
* Patients with hypersensitivity or allergy to the active pharmaceutical ingredient (API) or other ingredients used in the investigational drug, or patients with a history of severe allergy to other drugs (anaphylaxis, etc.).
* Patients with angle-closure glaucoma.
* Patients with disease or findings that are judged to affect this study from the viewpoint of safety and/or evaluation.
* Patients who received Levodopa-carbidopa continuous infusion gel therapy (LCIG therapy) or patients who plan to receive it during the study period.
* Patients who have used apomorphine subcutaneous injection 30 mg within 1 month prior to obtaining informed consent or patients who plan to use apomorphine during the study period.
* Patients who have undergone brain surgery for Parkinson's disease (pallidotomy, deep brain stimulation, etc.) or patients who plan to undergo such surgery during the study period.
* Patients who received or plan to receive transcranial magnetic stimulation therapy within 6 months prior to consent.
* Patients with a history or comorbidities of drug abuse or alcoholism.
* Patients with a history or comorbidities of mental illness (schizophrenia, psychotic depression, etc.). However, psychiatric symptoms associated with Parkinson's disease are excluded.
* Patients with overt dementia or Mini-Mental State Examination (MMSE) score less than 24 points.
* Patients with a history of suicidal ideation or attempted suicide within the past year or a history of present illness.
* Patients with a history of malignant syndrome caused by antiparkinsonian drugs.
* Patients with clinically problematic brain, cardiovascular, hematological, autoimmune, endocrine, cardiovascular, renal, gastrointestinal, or respiratory diseases (including infectious diseases) that are judged by the investigator to have the potential to affect the conduct of this study from the perspective of safety and other factors.
* Patients with any of the following laboratory test results from screening tests:

  * A creatinine level greater than or equal to 2 times the laboratory upper limit
  * Total bilirubin level greater than or equal to 3 times the laboratory upper limit
  * ALT or AST greater than or equal to 3 times the laboratory upper limit
  * ALP greater than or equal to 3 times the laboratory upper limit
* Patients who have clinically significant abnormalities in "other tests (including clinical tests)" in the screening test and are judged by the investigator to be inappropriate for participation in this study.
* Patients with acquired immunodeficiency syndrome (AIDS) (including patients who are either HIV antigen or antibody positive) or hepatitis (including patients who are HBs antigen positive or HCV antibody positive).
* Patients who required treatment for malignant tumors within 5 years before consent was obtained (excluding treated cervical intraepithelial neoplasia, cured nonmetastatic squamous or basal cell tumors of the skin).
* Patients who are scheduled for surgery requiring hospitalization during the study period or who are in a condition requiring surgery.
* Patients who are pregnant, breastfeeding, may be pregnant, or wish to become pregnant during the study period.
* Patients who have received all other unapproved drugs (including investigational drugs, drugs administered through clinical research, unapproved combination drugs, and new formulations) within 3 months prior to obtaining consent or within 5 times the half-life, whichever is longer.
* Patients who have received TR-012001 in the past.
* Patients who are deemed inappropriate for participation in this study by the investigator for any reason, including patients who have difficulty communicating or cooperating.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-09-28 (Actual); Primary Completion 2024-04-26 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Safety evaluation of TR-012001: Incidents of Treatment-Emergent Adverse Events | Day of administration of TR-012001/placebo (Day3) to the day of leaving the facility (Day4). If any adverse event(s) continue or occur on Day4, follow-up will be conducted until recovery or until the investigator decides no longer follow-up is necessary.
  Name of adverse event, date and time of onset, severity, seriousness, outcome, date and time of outcome, and relationship to TR-012001 of all adverse events (including serious adverse events) are evaluated.
Safety evaluation of TR-012001: Incidents of physical findings | 4 days and 3 nights
  The examination will include general findings and evaluation of the skin, eyes, ears/nose/throat, heart, chest, and abdomen. Record anything that is not normal, including those due to the subject's illness.
Safety evaluation of TR-012001: Vital sign (body temperature) | 4 days and 3 nights
  The results of vital signs will be used by the investigator to determine whether there are any safety issues continuing to participate in this study.
Safety evaluation of TR-012001: Vital sign (blood pressure) | 4 days and 3 nights
  The results of vital signs will be used by the investigator to determine whether there are any safety issues continuing to participate in this study. Blood pressure is measured in sitting state.
Safety evaluation of TR-012001: Vital sign (pulse rate) | 4 days and 3 nights
  The results of vital signs will be used by the investigator to determine whether there are any safety issues continuing to participate in this study. Pulse rate is measured in sitting state.
Safety evaluation of TR-012001: Columbia Suicide Severity Rating Scale (C-SSRS) | Day 1 and Day 4
  To evaluate the safety and tolerability of TR-012001, Columbia-Suicide Severity Rating Scale (C-SSRS) (Japanese version) is used to evaluates suicidal ideation and behavior.
  Scale range: Yes or No response to 11 questions, with minimum to maximum range of 0 to 5. Lower score represents better outcomes. Subscales not applicable.
Safety evaluation of TR-012001: Incidents of participants with laboratory abnormality | Day 1 and Day 4
  The results of laboratory test values (hematological, blood biochemical, and urinary tests) will be used by the investigator to determine whether there are any safety issues continuing to participate in this study.
Pharmacokinetics of TR-012001: Maximum plasma concentration (Cmax) | Pre-dose (baseline) and specified time points of post-dose
  Maximum observed plasma concentration of TR-012001.
Pharmacokinetics of TR-012001: Time to reach maximum plasma concentration (Tmax) | Pre-dose (baseline) and specified time points of post-dose
  Time to maximum observed plasma concentration of TR-012001.
Pharmacokinetics of TR-012001: Elimination half-life (t1/2) | Pre-dose (baseline) and specified time points of post-dose
  Elimination half-life.
Pharmacokinetics of TR-012001: Area under the plasma concentration-time curve (AUC0-inf) | Pre-dose (baseline) and specified time points of post-dose
  Area under the plasma concentration-time curve.
Pharmacokinetics of TR-012001: Mean residence time (MRT) | Pre-dose (baseline) and specified time points of post-dose
  Mean residence time.
Pharmacokinetics of TR-012001: Apparent whole body clearance (CL/f) | Pre-dose (baseline) and specified time points of post-dose
  Apparent whole body clearance.
Pharmacokinetics of TR-012001: Volume of distribution (Vd/f ) | Pre-dose (baseline) and specified time points of post-dose
  Volume of distribution.

CONTACTS AND LOCATIONS:
Overall Officials: Akihisa Mori, PhD, Study Director — SNLD, Ltd.
Locations (1):
- Saiseikai Imabari Hospital, Imabari, Ehime, Japan

IPD SHARING:
Plan to Share IPD: No